CLINICAL TRIAL: NCT00213330
Title: Cerebral Activity During Rectal Pain in Patients With Irritable Bowel Syndrome or Inflammatory Bowel Disease:Resonance Magnetic Imaging Study.
Brief Title: Cerebral Resonance Magnetic Imaging During Rectal Distention
Status: Withdrawn | Type: Observational
Why Stopped: patients with inflammatory colitis not included
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2001/105/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Ulcerative Colitis; Irritable Bowel Syndrome
Keywords: cerebral activity; rectal distension; colitis ulcerative; irritable bowel syndrome; magnetic resonance imaging
MeSH Terms: conditions — Colitis, Ulcerative; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: rectal distension

SUMMARY:
Irritable bowel syndrome is responsible for chronic abdominal pain, diarrhea and/or constipation. It is a very frequent problem. However, the exact cause of irritable bowel syndrome remains unknown. The purpose of this study is to look for a different cerebral response by magnetic resonance imaging after rectal stimulation in patients with irritable bowel syndrome compared to healthy subjects and to patients with digestive organic disease. Our hypothesis is that irritable bowel syndrome could be a problem of cerebral integration of visceral stimulation.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects irritable bowel syndrome (Rome II criteria) colitis ulcerative

Exclusion Criteria:

pregnant or breast feeding metallic material implanted good tolerance of rectal distension acute phase of ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects and patients with irritable bowel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-04; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Gérardin, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University hospital of Rouen, Rouen, France